CLINICAL TRIAL: NCT05111002
Title: Lefamulin for Mycoplasma Genitalium Treatment Failures in the US
Brief Title: Lefamulin for M. Genitalium Treatment Failures
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: At Sponsor Request
Sponsor: University of Washington (Other)
Collaborators: Nabriva Therapeutics AG (Industry)
Responsible Party: Principal Investigator, Lisa Manhart, Professor, Epidemiology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00012927
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Mycoplasma Genitalium Infection
Keywords: Lefamulin; Doxycycline; M. genitalium
MeSH Terms: interventions — lefamulin; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lefamulin alone (Experimental): Lefamulin 600mg tablet orally twice daily for 7 days
  Interventions: Drug: Lefamulin
- Doxycycline followed by lefamulin (Experimental): Doxycycline 100mg tablet orally twice daily for 7 days followed by lefamulin 600mg tablet orally twice daily for 7 days
  Interventions: Drug: Lefamulin; Drug: Doxycycline

INTERVENTIONS:
Drug: Lefamulin — 600mg tablet orally twice daily
  Other Names: Xenleta
Drug: Doxycycline — 100mg tablet orally twice daily
  Arms: Doxycycline followed by lefamulin

SUMMARY:
The purpose of this drug study is to find out whether the antibiotic lefamulin (trade name Xenleta) will cure Mycoplasma genitalium infections that have not been cured by prior antibiotics while finding out whether it is more effective if the antibiotic doxycycline is taken first.

DETAILED DESCRIPTION:
Study participants will be randomly chosen to receive either lefamulin alone or doxycycline followed by lefamulin in a 1:1 ratio. Each participant will receive 14 lefamulin pills or 14 doxycycline pills and 14 lefamulin pills in the mail and take them as directed for one week (each). Participants will collect one culture sample and one sample to confirm M. genitalium infection on the same day they take their first pill then mail the two samples to the laboratory. They will also answer questions about their symptoms, any side effects, and their behavior with their sex partners. Participants will collect samples two more times and answer questions three more times if they are randomly chosen to receive lefamulin alone or four more times if they are randomly chosen to receive doxycycline followed by lefamulin during the study. The study team will culture M. genitalium then determine minimum inhibitory concentrations (MICs) to three antibiotics (azithromycin, moxifloxacin, and lefamulin) to see whether it is resistant to any of these antibiotics. The study team will also test for M. genitalium to confirm whether the participants have an infection at baseline and see if lefamulin cured the infection upon completion of the lefamulin.

After 20 patients have been enrolled, the study team will conduct an interim analysis to assess futility. Futility will be defined as less than five percent probability that true efficacy is greater than or equal to 60 percent (i.e., less than or equal to three of the first 10 participants experience microbiologic cure). If neither lefamulin alone nor doxycycline followed by lefamulin meets criteria for futility, the study team will continue the study. If one regimen meets criteria for futility, the study team will drop the regimen that met the criteria for futility and continue to administer the other regimen to the remaining 20 participants. If both regimens meet criteria for futility, the study team will halt the study.

Study participants will be informed of their M. genitalium test of cure results. If the lefamulin does not cure the infection, the study physician will consult with the referring physician who will continue to treat the infection per clinic standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Physician referral
* Persistent symptomatic urogenital M. genitalium infection documented by any nucleic acid amplification test (NAAT) 14-90 days after completion of the prior antimicrobial regimen for M. genitalium
* Low risk of reinfection, defined as no unprotected sex with an untreated sex partner since completion of the prior antimicrobial regimen for M. genitalium
* Living in the United States
* Male or female sex at birth
* At least 18 years of age
* English-speaking
* Able to provide written informed consent
* Able to undergo a test to confirm M. genitalium infection at baseline and tests of cure 21-28 days and 42-47 days after completion of the lefamulin
* Referring physician willing and able to provide needed patient information

Exclusion Criteria:

* Rectal M. genitalium infection only
* Females with pelvic inflammatory disease (PID), pregnancy, or currently breastfeeding
* Females of reproductive age not on a highly effective method of contraception (i.e., intrauterine device (IUD), Nexplanon, progesterone only depot injection with last injection less than three months prior, oral contraceptive pill and last menstrual period less than 28 days prior)
* Known QT prolongation or ventricular arrhythmias including torsades de pointes
* Receiving concurrent drugs known to prolong QT interval (i.e., Class IA or III antiarrhythmics, antipsychotics, erythromycin, pimozide, moxifloxacin, tricyclic antidepressants)
* Receiving strong or moderate CYP3A or P-gp inducers, strong CYP3A or P-gp inhibitors, moderate CYP3A or P-gp inhibitors, or sensitive CYP3A4 substrates that prolong QT interval
* Moderate or severe liver impairment
* Known liver disease
* Renal failure requiring dialysis
* Known allergy to doxycycline, other tetracyclines, and/or lefamulin
* Unwilling or unable to undergo a test to confirm M. genitalium infection at baseline or tests of cure 21-28 days and 42-47 days after completion of the lefamulin
* Not fluent in English and/or not able to provide written informed consent
* Referring physician unwilling or unable to provide needed patient information
* At the study physician's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa E Manhart, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Not federally funded. Currently no IPD sharing plan.

RESULTS

PARTICIPANT FLOW:
Period: Primary Outcome
Arm/Group | Lefamulin Alone | Doxycycline Followed by Lefamulin
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Negative Confirmatory Aptima MG Test | 1 | 0
Period: Secondary Outcome
Arm/Group | Lefamulin Alone | Doxycycline Followed by Lefamulin
Started | 5 | 6
Completed | 4 | 6
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lefamulin Alone | Doxycycline Followed by Lefamulin | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [33 to 39] | 40 [34 to 44] | 39 [33 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 1 | 4 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Confirmatory MG Test [Count of Participants; unit: Participants] — Confirmatory Aptima Mycoplasma genitalium test
  Participants
    Positive | 5 | 6 | 11
    Negative | 1 | 0 | 1
    Indeterminate | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Microbiologic Cure
Description: Defined as a negative Aptima Mycoplasma genitalium test 21-28 days after completion of the lefamulin
Time Frame: 21-28 days after completion of the lefamulin
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lefamulin Alone | Doxycycline Followed by Lefamulin
Number analyzed (Participants) | 5 | 6
percentage of participants | 60 [15 to 95] | 50 [12 to 88]

2. Secondary Outcome: Number and Percentage of Participants With Sustained Microbiologic Cure
Description: Defined as a negative Aptima Mycoplasma genitalium test 42-47 days after completion of the lefamulin
Time Frame: 42-47 days after completion of the lefamulin
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lefamulin Alone | Doxycycline Followed by Lefamulin
Number analyzed (Participants) | 4 | 6
percentage of participants | 50 [7 to 93] | 50 [12 to 88]

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Lefamulin Alone | Doxycycline Followed by Lefamulin
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 5/5 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Lefamulin Alone (N=5) | Doxycycline Followed by Lefamulin (N=6)
Nausea (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 4
Sensitivity to Light (Skin and subcutaneous tissue disorders) | 0/0 | 1
Vaginal Yeast Infection (Infections and infestations) | 0/0 | 0
Other (General disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
This trial was stopped early due to cessation of operations by the antibiotic manufacturer and expiration of study drug. The number of study participants was less than designed and the small number of people resulted in unstable efficacy estimates and wide 95% confidence intervals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT05111002/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT05111002/ICF_001.pdf